CLINICAL TRIAL: NCT01523249
Title: Three-Dimensional Ultrasound (3D US) for Epidural Needle Insertion in Parturients
Brief Title: Three-Dimensional Ultrasound (3D US) in Parturients
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: H10-01974
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Pregnancy
Keywords: 3D ultrasonography; epidural; neuraxial anesthesia; neuraxial analgesia; pregnant woman; parturients
MeSH Terms: interventions — Palpation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Scanned and palpated: Healthy, pregnant, term women delivering at BC Women's Hospital and expecting to have neuraxial anesthesia.
  Interventions: Device: Lumbar 3D ultrasound scanning and palpation (Ultrasonix )

INTERVENTIONS:
Device: Lumbar 3D ultrasound scanning and palpation (Ultrasonix ) — Paramedian ultrasound scanning of L2-3 and L3-4 lumbar interspaces to visualize ligamentum flavum. Palpation of the same intervertebral spaces to identify spine midline and needle insertion point.
  Other Names: Ultrasonix US machine (model Sonix Touch)

SUMMARY:
The purpose of this study is to compare accuracy of a new three-dimensional ultrasound (3D US) technique with the traditional palpation method for identification of the needle insertion site on patients' skin before epidural needle placement in pregnant women. The investigators hypothesize that the needle puncture site identified by 3D US is located within a 5 mm radius from the puncture site identified by palpation.

DETAILED DESCRIPTION:
Traditionally, the manual palpation of lower back is used to identify the skin insertion point for the epidural needle placement in obstetric patients. Recently, two-dimensional ultrasound (2D US) scanning before the epidural needle insertion proved to improve an accurate determination of inter-vertebral levels and spine midline. 2D US is also useful in determining the depth to the epidural space and needle insertion angle. A three-dimensional ultrasound (3D US) technique is a new advancement in the ultrasound technology. 3D US allows for a real-time, visual guidance of the epidural needle insertion. This study will assess weather 3D US, compared to palpation, can accurately identify the skin needle insertion site for the epidural needle placement.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Greater than or equal to 19 years old
* Term pregnancy (greater than or equal to 38 weeks gestation age)
* Ability to read English in order to understand the consent form

Exclusion Criteria:

* BMI greater than or equal to 40
* Scoliosis
* Previous difficult regional anesthesia/analgesia
* Previous lower back surgery
* Active labour
* Allergy to epidural tape, surgical paper tape, or felt pen

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Term pregnant women expecting neuraxial anesthesia or analgesia for cesarean delivery or labour pain control at BC Women's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Distance between two needle insertion points | 20 minutes of testing prior to delivery
  To measure the distance between the needle puncture site identified by the 3D US transducer to the needle puncture site identified by palpation, measured on a transparency film.

SECONDARY OUTCOMES:
Distance between needle insertion point and spine midline | 20 minutes of testing prior to delivery
  To measure the perpendicular distance between the needle puncture site identified by the 3D US transducer to the midline identified by manual palpation (to the P-line), measured on a transparency film.
assess quality of 3D US images | one year
  To obtain US images of the epidural anatomy with various settings of the image-processing system to determine the optimal 3D US parameters that give the clearest images. An experienced sonographer will analyze the US images in the UBC laboratory using a qualitative measure of clarity (scale of 1 to 5) of the depiction of the ligamentum flavum and laminae. This quality measure will be correlated to the image acquisition parameters to determine the optimal set of parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Allaudin Kamani, MD, Principal Investigator — University of British Columbia and BC Women's Hospital
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada